CLINICAL TRIAL: NCT02473887
Title: Flavored Intravenous Ondansetron Administered Orally for the Treatment of Persistent Vomiting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00030
Record Dates: First submitted 2015-05-25; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-05

CONDITIONS: Gastroenteritis
Keywords: ondansetron; palatability; vomiting
MeSH Terms: conditions — Gastroenteritis; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gastroenteritis with persistent vomiting. (Experimental): patients with gastroenteritis with persistent vomiting received single dose of intravenous ondansetron form orally after being flavored with 1:1 ORA-sweet, the dose of ondansetron was determined based on the patient presenting weight.
  Interventions: Drug: Ondansetron with1:1 ORA - sweet.

INTERVENTIONS:
Drug: Ondansetron with1:1 ORA - sweet. — single dose of intravenous ondansetron form orally after being flavored with 1:1 ORA-sweet, the dose of ondansetron was determined based on the patient presenting weight.
  Other Names: Zofran

SUMMARY:
The purpose of this study is to give children with gastroenteritis with persistent vomiting flavored intravenous ondansetron orally. The investigators test the palatability of the drug and check the serum level of ondansetron at 4 hours .

DETAILED DESCRIPTION:
This is a prospective pilot study for children,3-8 years of age presented to the Pediatric Emergency Department in the state of Qatar between September 2014 and January 2015, with acute gastroenteritis with mild to moderate dehydration, more than 2 episodes of vomiting in the last 24 hours, and who had failed oral rehydration trial in the department as per the department oral hydration protocol. Acute gastroenteritis was defined as diarrhea and vomiting for less than a week period.

Hydration level was assessed for all patients on arrival, and eligible patients were enrolled after obtaining an informed written consent.Enrolled patients received intravenous ondansetron form orally after being flavored 1:1 with ORA-sweet, the dose of ondansetron was determined based on the patient presenting weight. Palatability was evaluated by the primary investigator within one minute fom drug administration applying taste scores for children and recorded according to a specific scoring system. All patients were kept nil per oral for 30 minutes and then oral rehydration trial was started as per the department rehydration protocol. If the drug was vomited within 30 min of administration, a similar second dose was given. Blood level for ondansetron was collected 4 hours after the successful drug administration and was sent to the department laboratory within 5 min. Patients were sent home when they were ready for discharge as per the treating physician discretion. All patients were followed by a telephone call after 24 hours to assess the safety and efficacy of the orally taken ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* children 3-8 years of age.
* acute simple gastroenteritis with mild to moderate dehydration.
* more than 2 episodes of vomiting in 24 hours period.

Exclusion Criteria:

* known hypersensitivity to ondansetron.
* seizure disorder.
* chronic liver or kidney diseases.
* on any chronic medication.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
ondansetron serum level. | 4 hour
  serum level of ondansetron at 4 hours after drug administration.

SECONDARY OUTCOMES:
palatability score of the drug.score 3/5( not sure to like very much ). | within one minute from drug administration.
  Palatability was evaluated by the primary investigator within one minute fom drug administration applying taste scores for children and recorded according to a specific scoring system. score 3/5( not sure to like very much ).

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Al-Ansari, MD, FRCPC, FAAP, Study Chair — Hamad Medical Corporation, Doha - Qatar

REFERENCES:
- [Background] Freedman SB, Adler M, Seshadri R, Powell EC. Oral ondansetron for gastroenteritis in a pediatric emergency department. N Engl J Med. 2006 Apr 20;354(16):1698-705. doi: 10.1056/NEJMoa055119. PMID 16625009
- [Background] DeCamp LR, Byerley JS, Doshi N, Steiner MJ. Use of antiemetic agents in acute gastroenteritis: a systematic review and meta-analysis. Arch Pediatr Adolesc Med. 2008 Sep;162(9):858-65. doi: 10.1001/archpedi.162.9.858. PMID 18762604
- [Background] Sturm JJ, Pierzchala A, Simon HK, Hirsh DA. Ondansetron use in the pediatric emergency room for diagnoses other than acute gastroenteritis. Pediatr Emerg Care. 2012 Mar;28(3):247-50. doi: 10.1097/PEC.0b013e3182494d87. PMID 22344213
- [Background] Angelilli ML, Toscani M, Matsui DM, Rieder MJ. Palatability of oral antibiotics among children in an urban primary care center. Arch Pediatr Adolesc Med. 2000 Mar;154(3):267-70. doi: 10.1001/archpedi.154.3.267. PMID 10710025